CLINICAL TRIAL: NCT05143268
Title: Impact of Acupuncture on Acute Dysphagia in Patients Treated With Radio-chemotherapy for Head and Neck Squamous Cell Carcinoma: a Randomized Phase 2 Study
Brief Title: Acupuncture for Dysphagia in Head and Neck Squamous Cell Carcinoma
Acronym: ACP-HN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lorenzo Livi (Other)
Responsible Party: Sponsor-Investigator, Lorenzo Livi, Professor, Azienda Ospedaliero-Universitaria Careggi
Organization: Azienda Ospedaliero-Universitaria Careggi (Other)
Other Study IDs: ACP-HN
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: In the experimental arm (arm A), a total of 11 sessions of acupuncture will be performed on a weekly basis, spanning from 2 weeks before Radiotherapy start throughout 7 weeks of treatment, to 2 weeks after its completion. Patients randomized to the experimental arm will receive acupuncture in addition to standard of care treatment, chosen by the treating multidisciplinary team in accordance with international guidelines.
- B: In the standard arm (arm B), patients will be treated with standard of care treatment.

SUMMARY:
This is a randomized phase 2 study on the impact of acupuncture on acute dysphagia in patients treated with radio-chemotherapy for head and neck squamous cell carcinoma

DETAILED DESCRIPTION:
In order to attempt to reduce the impact of adverse effects produced by oncological treatments, cancer patients frequently turn to complementary integrative therapies.

Among them, acupuncture has been characterized by a growing role in cancer-related symptoms management in last 10 years.

After FDA approval for use as a medical device in 1996, the application of this technique in oncology has been on the rise in the Western countries.

By modulating brain regions involved in cognition and emotion, some degree of successful symptom management with acupuncture has been demonstrated in oncology In the context of head and neck cancer, the first application of acupuncture was related to chronic shoulder pain and dysfunction following neck dissection.

The primary objective of the study is to compare the effect of acupuncture and standard treatment on swallowing function assessed with MDADI scale (MD Anderson Dysphagia Inventory) 2 weeks after the end of RT (end of treatment, EoT).

ELIGIBILITY:
Inclusion Criteria:

* histologically-confirmed diagnosis of squamous cell carcinoma of the nasopharynx, oropharynx, hypopharynx and larynx or histologically-confirmed diagnosis of undifferentiated carcinoma of the nasopharynx
* by judgement of the local investigator, indication for a DNST with curative intent, consisting of one of the 3 following options:

  * radiotherapy alone
  * cisplatin-based concomitant chemo-radiotherapy
  * cetuximab-based concomitant bio-radiotherapy
* clinical stage of disease: II, III, IVA, IVB (according to TNM/AJCC 8th edition) for primary tumors of the larynx, hypopharynx and oropharynx (p16/HPV negative), provided that for stage II disease (cT2N0) the local investigator will prescribe an elective irradiation of regional lymph nodes
* clinical stage of disease: I, II, III (according to TNM/AJCC 8th edition) for primary tumors of the oropharynx (p16/HPV positive), provided that for stage I disease (cT1N0) the local investigator will prescribe an elective irradiation of regional lymph nodes

Exclusion Criteria:

* histologically-confirmed head and neck cancer of any other primary anatomic location in the head and neck not specified in the inclusion criteria including patients with HNSCC of unknown primary or non-squamous histologies
* metastatic disease
* gross total excision of both primary and nodal disease before index treatment
* surgical manipulation including therapeutic tonsillectomy, local excision of primary site, and nodal excision that removes all clinically and radiographically evident disease
* prior radiotherapy to the head and neck region
* induction chemotherapy prior to radiotherapy
* prior use of acupuncture for SCCHN or for different indications
* prior allergic reaction or history of hypersensitivity to inox austenitic steel (Cr18Ni9)
* active or prior documented neurologic or rheumatologic disorder with a potential impact on the swallowing function (i.e: multiple sclerosis, amyotrophic lateral sclerosis, scleroderma)
* active process of severe skin infection in the neck contraindicating the execution of acupuncture in the opinion of the investigator
* severe baseline dysphagia documented by a MDADI scale (MD Anderson Dysphagia Inventory) composite score below 60
* any condition that, in the opinion of the investigator, would not require to encompass at least ipsilateral neck lymph nodes in the irradiation field
* any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over 18 years old who have received a histologically-confirmed diagnosis of squamous cell carcinoma of the nasopharynx, oropharynx, hypopharynx and larynx or histologically-confirmed diagnosis of undifferentiated carcinoma of the nasopharynx
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-06-03 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Primary objective | two weeks after the end of treatment
  Swallowing function assessed with MDADI scale (MD Anderson Dysphagia Inventory)

SECONDARY OUTCOMES:
Secondary objective n.1 | 12 weeks after end of treatment
  Swallowing function assessed with MDADI scale (MD Anderson Dysphagia Inventory)
Secondary objective n.2 | 24 weeks after end of treatment
  Swallowing function assessed with MDADI scale (MD Anderson Dysphagia Inventory)
Secondary objective n.3 | 12 and 24 weeks after end of treatment
  Patients' quality of life assessed with the EORTC QLQ-C30 and QLC-HN 43
Secondary objective n.4 | maximum of 11 weekly sessions
  Feasibility of acupuncture (percentage of completed acupuncture sessions out of planned per protocol)
Secondary objective n.5 | 2 weeks after end of treatment
  Incidence of moderate-severe dysphagia (>G2) assessed with CTCAE v. 5.0
Secondary objective n.6 | 2 weeks after end of treatment
  Incidence of moderate-severe adverse events (G3-G4) assessed with CTCAE v.5
Secondary objective n.7 | 2 weeks after the end of treatment
  Relative dose intensity of systemic therapy
Secondary objective n.8 | 2 weeks after end of treatment
  Radiation interruptions
Secondary objective n.9 | 2 weeks after end of treatment
  Relative weight loss (percentage of weight loss compared with baseline value at start of therapy)

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - AOU Careggi Radiation Oncology Unit, Florence
  - Azienda Ospedaliero Universitaria Careggi, Florence